CLINICAL TRIAL: NCT03876028
Title: A Phase Ib, Multicenter Study to Determine the Safety and Tolerability of Tisagenlecleucel in Combination With Ibrutinib in Adult Patients With Relapsed and/or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Study of Tisagenlecleucel in Combination With Ibrutinib in r/r Diffuse Large B-cell Lymphoma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019L12101C
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma; Diffuse Large B-cell lymphoma; DLBCL; r/r Diffuse Large B-cell Lymphoma; relapsed/refractory DLBCL; CTL019; Tisagenlecleucel; Ibrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence | interventions — tisagenlecleucel; ibrutinib

STUDY DESIGN:
Intervention Model Description: "The study will enroll patients into two arms in parallel: Arm 1: Patients will start ibrutinib treatment before leukapheresis. Arm 2: Patients will start ibrutinib treatment after leukapheresis. Approximately 3-6 patients will be enrolled into each of the two arms in parallel. An early safety review will be performed after these patients have received sufficient ibrutinib treatment and tisagenlecleucel infusion, and have completed at least 21 days of follow up. Additional patients (up to 20 total) will be enrolled into both arms to further characterize the safety, tolerability and preliminary efficacy of ibrutinib in combination with tisagenlecleucel."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrutinib (before leukapheresis) + Tisagenlecleucel (Experimental): Patients will start ibrutinib treatment before leukapheresis
  Interventions: Biological: Tisagenlecleucel; Drug: Ibrutinib
- Ibrutinib (after leukapheresis) + Tisagenlecleucel (Experimental): Patients will start ibrutinib treatment after leukapheresis.
  Interventions: Biological: Tisagenlecleucel; Drug: Ibrutinib

INTERVENTIONS:
Biological: Tisagenlecleucel — Infusion
Drug: Ibrutinib — Oral (tablets or capsules)

SUMMARY:
A multi-center, open-label, phase Ib study to evaluate the safety and tolerability of the administration of tisagenlecleucel in combination with ibrutinib in patients with r/r DLBCL who have received two or more lines of systemic therapy, including an anti-CD20 and anthracycline based chemotherapy, and who have progressed after or are not candidates for ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed DLBCL as per the local histopathological assessment.
2. Relapsed or refractory disease having received 2 or more lines of systemic therapy, including anti-CD20 and anthracycline based chemotherapy, and either having progressed after (or relapsed after) ASCT, or being ineligible for or not consenting to ASCT.
3. Measurable disease at time of enrollment.
4. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening.
5. Adequate renal, liver, and bone marrow, organ function, and minimum level of pulmonary reserve.

Exclusion Criteria:

1. Patients with Richter's transformation, Burkitt's lymphoma, and primary DLBCL of the CNS.
2. Prior anti-CD19 directed therapy.
3. Prior gene therapy.
4. Prior adoptive T cell therapy.
5. Prior ibrutinib therapy within the 30 days prior to screening.
6. Patients with active CNS involvement are excluded, except if the CNS involvement has been effectively treated and provided that local treatment was > 4 weeks before enrollment.
7. Prior allogeneic HSCT
8. . Significant cardiac abnormality including history of myocardial infarction within 6 months prior to screening as detailed in the study protocol.

Other eligibility criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 24 months
  Month 24 is planned study end
Severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months
  Month 24 is planned study end
Ibrutinib dose modification following tisagenlecleucel infusion | 24 months
  Month 24 is planned study end

SECONDARY OUTCOMES:
Response Rate | Month 3
  3-months post tisagenlecleucel infusion, assessed by local investigator according to Lugano criteria
Response Rate | Month 6
  6-month post tisagenlecleucel infusion, assessed by local investigator according to Lugano criteria
Overall Response Rate | 24 months
Duration of Response | 24 months
Progression Free Survival (PFS) | 24 months
Overall Survival (OS) | 24 months
Tisagenlecleucel transgene concentrations | 24 months
  qPCR will be used to measure tisagenlecleucel transgene concentrations in available tissue, such as peripheral blood, bone marrow, tumor/lymph node tissue, and/or CSF.
Cellular kinetics of Tisagenlecleucel (Cmax) | 24 months
  Cmax cellular kinetics parameter (via qPCR) for tisagenlecleucel in the presence of ibrutinib
Cellular kinetics of Tisagenlecleucel (Tmax) | 24 months
  Tmax cellular kinetics parameter (via qPCR) for tisagenlecleucel in the presence of ibrutinib
Cellular kinetics of Tisagenlecleucel (AUC) | 24 months
  AUC cellular kinetics parameter (via qPCR) for tisagenlecleucel in the presence of ibrutinib
Cellular kinetics of Tisagenlecleucel (Clast) | 24 month
  Clast cellular kinetics parameter (via qPCR) for tisagenlecleucel in the presence of ibrutinib
Cellular kinetics of Tisagenlecleucel (Tlast) | 24 month
  Tlast cellular kinetics parameter (via qPCR) for tisagenlecleucel in the presence of ibrutinib
Anti-drug antibody (ADA) response to Tisagenlecleucel (humoral immunogenicity) | 24 months
  Pre-existing and treatment related immunogenicity (humoral) of tisagenlecleucel will be characterized by flow cytometry
Anti- tisagenlecleucel t-cell response (cellular immunogenicity) | 24 months
  Pre-existing and treatment related immunogenicity (cellular) of tisagenlecleucel will be characterized IFN-g staining and flow cytometry
Characterize cellular kinetic parameters in the presence of ADA and/or anti-tisagenlecleucel t-cell response | 24 months
Characterize efficacy of tisagenlecleucel in the presence of ADA and/or anti-tisagenlecleucel t-cell response | 24 month

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Chavez JC, Napier E, Bondanza A, Lewandowski A, Mataraza J, Quinn D, Kwon P, Locke FL, Engels B, Awasthi R, Georgala P, Leyk M, Hynds D, Moschetta M, Schuster SJ. Tisagenlecleucel in combination with ibrutinib in adults with relapsed and/or refractory large B-cell lymphomas. Blood Neoplasia. 2025 Oct 24;3(1):100176. doi: 10.1016/j.bneo.2025.100176. eCollection 2026 Feb. PMID 41536778
- See also: Study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17966
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1223